CLINICAL TRIAL: NCT05881486
Title: The Effects of Intravenous Fosaprepitant and Ondansetron for the Prevention of Postoperative Nausea and Vomiting in Thoracicsurgery Patients: A Single-center, Randomized, Double-Blinded Clinical Study
Brief Title: Antiemetic Prophylaxis With Fosaprepitant and Ondansetron in Patients Undergoing Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYLL-202210-072-1
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Nausea and Vomiting; Anesthesia Complication; Thoracic Diseases
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Thoracic Diseases | interventions — Ondansetron; fosaprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fosaprepitant (Experimental): Participants undergoing thoracoscopic pneumonectomy will receive 150 mg of fosaprepitant and 100 ml of normal saline, administer intravenously after the induction of general anesthesia.
  Interventions: Drug: Fosaprepitant 150 mg
- Ondansetron (Active Comparator): Participants undergoing thoracoscopic pneumonectomy received 8 mg of ondansetron and 100 ml of normal saline, administer intravenously after the induction of general anesthesia.
  Interventions: Drug: Ondansetron 8mg

INTERVENTIONS:
Drug: Ondansetron 8mg — 8 mg Ondansetron+100 ml normal saline
  Arms: Ondansetron
Drug: Fosaprepitant 150 mg — 150 mg fosaprepitant +100 ml normal saline
  Arms: Fosaprepitant

SUMMARY:
The goal of this clinical trial is to compare the efficacy, safety and feasibility of intravenous Fosaprepitant and Ondansetron for the prevention of postoperative nausea and vomiting in thoracicsurgery patients. Participants will be randomized in a 1:1 ratio to the Fosaprepitant and Ondansetron group.The groups were analyzed and compared for frequency of vomiting in 24 h after surgery. In addition, we will further compare the occurrence of postoperative pulmonary complications, length of hospital stay, nutrition and quality of life after surgery in patients treated with different antiemetic prophylaxis.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common postoperative complication of general anesthesia. The antiemetic 5-serotonin 3 (5-HT 3) receptor antagonist is widely used in postoperative anti-emesis,However, more clinical studies are needed to confirm whether neurokinin-1 (NK-1) receptor antagonists have better effects on PONV than 5-HT 3 receptor antagonists.We aimed to evaluate the effects of NK-1 receptor antagonists and 5-HT 3 receptor antagonists on PONV through a randomized controlled study. To this end, we took patients undergoing thoracic surgery as the research object, they received an antiemetic prophylaxis with ondansetron or fosaprepitant, and the frequency of postoperative nausea and vomiting the of the two antiemetic prophylaxis regimens were analyzed, and the occurrence of pulmonary complications, length of hospital stay, the nutrition and quality of life after surgery administration were also compared. Through this clinical trial, we hope to obtain a better antiemetic prophylaxis regimen and provide clear information for patients and physicians to guide clinical decisions that enhance treatment efficacy and reduce the occurrence of side effects.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 70 years
2. physical status classified by the American Society of Anesthesiologists (ASA) scale as I to III
3. Apfel score ≥ 2
4. undergoing thoracoscopic pneumonectomy

Exclusion Criteria:

1. Preoperative disorders of consciousness
2. body mass index (BMI) > 35 kg/m2
3. occurrence of episodes of nausea or vomiting within 24 h prior to surgery、motion sickness,、previous PONV、people who smoke、people with alcoholism、use of corticosteroids, psychoactive or antiemetic drugs,、hypersensitivity to the study medications
4. serious kidney, liver, lung, heart, brain or bone marrow disease
5. conversion from thoracoscopic pneumonectomy to conventional pneumonectomy
6. participation in another clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of PONV within 24 hours | Day 1
  The groups will be analyzed and compared for frequency of nausea and vomiting in 24 h after surgery

SECONDARY OUTCOMES:
Incidence of PONV within 48 hours | Day 2
  The groups will be analyzed and compared for frequency of nausea and vomiting in 48 h after surgery
occurrence of Drug-related adverse effects | Day 3
  The groups will be compared for the incidence of unwanted effects of antiemetic medicines include onstipation,weakness, headache, dizziness and sleepiness.
Postoperative pain score | Day 3
  This project will be measured by patients' postoperative pain score.
The dosage of opioids used after surgery | Day 3
  This project will be measured by the dosage of opioid drugs used after surgery.
the length of hospital stay | From date of admission until the date of discharge, assessed up to 7 days.
  The groups will be compared for the time from admission to discharge
postoperative pulmonary complications | Day 3
  Postoperative pulmonary complications include respiratory infection,respiratory failure,pleural effusion,atelectasis and pneumothorax

REFERENCES:
- [Background] Apfel CC, Kranke P, Katz MH, Goepfert C, Papenfuss T, Rauch S, Heineck R, Greim CA, Roewer N. Volatile anaesthetics may be the main cause of early but not delayed postoperative vomiting: a randomized controlled trial of factorial design. Br J Anaesth. 2002 May;88(5):659-68. doi: 10.1093/bja/88.5.659. PMID 12067003
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Gan T, Sloan F, Dear Gde L, El-Moalem HE, Lubarsky DA. How much are patients willing to pay to avoid postoperative nausea and vomiting? Anesth Analg. 2001 Feb;92(2):393-400. doi: 10.1097/00000539-200102000-00022. PMID 11159239
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Dorman RB, Miller CJ, Leslie DB, Serrot FJ, Slusarek B, Buchwald H, Connett JE, Ikramuddin S. Risk for hospital readmission following bariatric surgery. PLoS One. 2012;7(3):e32506. doi: 10.1371/journal.pone.0032506. Epub 2012 Mar 7. PMID 22412881
- [Background] Parra-Sanchez I, Abdallah R, You J, Fu AZ, Grady M, Cummings K 3rd, Apfel C, Sessler DI. A time-motion economic analysis of postoperative nausea and vomiting in ambulatory surgery. Can J Anaesth. 2012 Apr;59(4):366-75. doi: 10.1007/s12630-011-9660-x. Epub 2012 Jan 6. PMID 22223185
- [Background] Andreae MH, Gabry JS, Goodrich B, White RS, Hall C. Antiemetic Prophylaxis as a Marker of Health Care Disparities in the National Anesthesia Clinical Outcomes Registry. Anesth Analg. 2018 Feb;126(2):588-599. doi: 10.1213/ANE.0000000000002582. PMID 29116968
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Bailey PL, Streisand JB, Pace NL, Bubbers SJ, East KA, Mulder S, Stanley TH. Transdermal scopolamine reduces nausea and vomiting after outpatient laparoscopy. Anesthesiology. 1990 Jun;72(6):977-80. doi: 10.1097/00000542-199006000-00005. PMID 2140929
- [Background] Gan TJ, El-Molem H, Ray J, Glass PS. Patient-controlled antiemesis: a randomized, double-blind comparison of two doses of propofol versus placebo. Anesthesiology. 1999 Jun;90(6):1564-70. doi: 10.1097/00000542-199906000-00011. PMID 10360853
- [Background] Navari RM, Aapro M. Antiemetic Prophylaxis for Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Apr 7;374(14):1356-67. doi: 10.1056/NEJMra1515442. No abstract available. PMID 27050207
- [Background] Hesketh PJ, Van Belle S, Aapro M, Tattersall FD, Naylor RJ, Hargreaves R, Carides AD, Evans JK, Horgan KJ. Differential involvement of neurotransmitters through the time course of cisplatin-induced emesis as revealed by therapy with specific receptor antagonists. Eur J Cancer. 2003 May;39(8):1074-80. doi: 10.1016/s0959-8049(02)00674-3. PMID 12736106
- [Background] Hata A, Okamoto I, Inui N, Okada M, Morise M, Akiyoshi K, Takeda M, Watanabe Y, Sugawara S, Shinagawa N, Kubota K, Saeki T, Tamura T. Randomized, Double-Blind, Phase III Study of Fosnetupitant Versus Fosaprepitant for Prevention of Highly Emetogenic Chemotherapy-Induced Nausea and Vomiting: CONSOLE. J Clin Oncol. 2022 Jan 10;40(2):180-188. doi: 10.1200/JCO.21.01315. Epub 2021 Nov 18. PMID 34793245
- [Background] Horn CC, Wallisch WJ, Homanics GE, Williams JP. Pathophysiological and neurochemical mechanisms of postoperative nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:55-66. doi: 10.1016/j.ejphar.2013.10.037. Epub 2013 Oct 26. PMID 24495419
- [Background] Murakami C, Kakuta N, Kume K, Sakai Y, Kasai A, Oyama T, Tanaka K, Tsutsumi YM. A Comparison of Fosaprepitant and Ondansetron for Preventing Postoperative Nausea and Vomiting in Moderate to High Risk Patients: A Retrospective Database Analysis. Biomed Res Int. 2017;2017:5703528. doi: 10.1155/2017/5703528. Epub 2017 Dec 19. PMID 29410964
- [Background] Weibel S, Rucker G, Eberhart LH, Pace NL, Hartl HM, Jordan OL, Mayer D, Riemer M, Schaefer MS, Raj D, Backhaus I, Helf A, Schlesinger T, Kienbaum P, Kranke P. Drugs for preventing postoperative nausea and vomiting in adults after general anaesthesia: a network meta-analysis. Cochrane Database Syst Rev. 2020 Oct 19;10(10):CD012859. doi: 10.1002/14651858.CD012859.pub2. PMID 33075160